CLINICAL TRIAL: NCT06701916
Title: Effect of a Person-centred Care Intervention on the Social Dimension of People With Chronic Heart Failure: A Randomised Controlled Trial
Brief Title: SHARE Study: Social Chronic Heart Failure Person-centred cARE Intervention
Acronym: SHARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: University of Navarra (Other); Hospital of Navarra (Other); University of Gothenburg Center for Person-Centred Care, GPCC (Unknown); Hospital Donostia (Other); Instituto de InvestigaciÃ³n Sanitaria de Navarra (IdiSNA) (Unknown)
Responsible Party: Principal Investigator, Maddi Olano, Associate Professor, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UNAV-SHARE
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
Keywords: Person-centredness; RCT; Process evaluation; Health plan; Partnership; Person-centred care; Person-centered care; patient-centered care; Heart failure; social isolation; social support; social dimension
MeSH Terms: conditions — Heart Failure; Social Isolation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment An RCT: Heart failure patients who consent to participate and meet the inclusion criteria will be randomized. Randomization will be conducted by research nurses. Participants will be randomly assigned to either the control or intervention group with a 1:1 allocation, according to computer-generated randomization. The control group will receive usual care, while the intervention group will receive a person-centered care intervention for three months in addition to usual care.
Masking Description: The nature of the intervention means that neither participants nor the health care professionals in the SHARE intervention can be blinded to allocation in the RCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Usual Care. Participants allocated to the control group will not receive any additional intervention. They will receive standard care for the outpatient management of their Heart Failure, based on the recommendations of the European Society of Cardiology guidelines for the follow-up of heart failure patients.
- Intervention group. (Experimental): The Person-Centred Care intervention will be delivered for 3 months on top of usual care.
  Interventions: Behavioral: Intervention group.; Behavioral: Usual care

INTERVENTIONS:
Behavioral: Intervention group. — The intervention will be carried out by a multidisciplinary team composed of nurses, doctors, social workers, and psychologists from each hospital. Through this intervention, a narrative from the patients will be obtained regarding their goals, desires, capabilities, and resources related to their health situation. A health plan will be jointly created, reflecting both short- and long-term objectives, identifying the resources available to the person and within their immediate environment, and outlining how they want and expect to receive support from healthcare professionals.
  Arms: Intervention group.
Behavioral: Usual care — Usual care for the outpatient management of Chronic Heart Failure.
  Arms: Intervention group.

SUMMARY:
People with Chronic Heart Failure (CHF) live with a complex situation that significantly affects their quality of life and well-being. Among the consequences of CHF that have the greatest impact on individuals is the effect it has on their social dimension. The symptomatic burden they experience, along with the influence of social determinants, social support, and psychosocial factors, results in disability and limitations in maintaining an adequate social life and roles, participating in social events, and having relationships beyond their closest family circle. Various international health organizations have emphasized the need to move towards Person-Centered Care (PCC). Adopting this approach involves shifting from a model in which the patient is a passive subject of a medical intervention to one in which the patient takes an active role in their care and decision-making process. The aim of this study is to assess the effectiveness of a PCC intervention on the social dimension of people with CHF. The study will be conducted at the Outpatient Heart Failure Units of Donostia University Hospital, the University Hospital of Navarra, and the University of Navarra Clinic in Pamplona. A randomized controlled, open-label, parallel-group, multicenter clinical trial will be carried out, based on the Medical Research Council framework. This will evaluate the effect of a three-month intervention consisting of in-person and telephone support centered on the person, in addition to usual care, compared to usual care alone, in a sample of 374 individuals. The intervention will be implemented by a multidisciplinary team comprising nurses, doctors, social workers, and psychologists from each hospital. Through this intervention, a patient narrative will be obtained regarding their goals, desires, capabilities, and resources related to their health situation. A health plan will be jointly created that will reflect short- and long-term goals, identify the resources available to the person and in their immediate environment, and outline how they want and expect to receive support from healthcare professionals. To assess its impact, the intervention's effect on the ability to participate in social roles and activities, perceived level of social isolation, and perception of social support will be measured. Additionally, the effect on self-efficacy perception, level of self-care and treatment adherence, anxiety and depression, and overall health experience with the disease will be evaluated, as well as rates of hospitalization, disease decompensation, emergency visits, and death.

DETAILED DESCRIPTION:
Background According to the WHO, heart disease has been the leading cause of mortality worldwide for the past 20 years. Specifically, people with Chronic Heart Failure (CHF) have become a priority group in healthcare systems. The prevalence of CHF in the adult population of industrialized countries reaches 3% and is expected to increase due to its chronic and progressive nature, driven by advances in healthcare. Currently, women make up 50.3% of the global prevalence, and it has been found that more than 10% of people over 70 suffer from it.

Several studies have shown that people with CHF live in a complex situation that significantly impacts their quality of life and overall well-being. This is because, on one hand, they must cope with complex treatment regimens, strict self-care behaviors, and lifestyle changes that affect their daily lives. On the other hand, they experience situations that lead to profound changes in all their personal dimensions, including physical restrictions, emotional and spiritual needs, and the impact on family and social roles. Despite this, the healthcare provided to these patients, as is the case with other chronic conditions, primarily focuses on disease management and the prevention of complications, while other aspects related to the experience of living with CHF are not being addressed.

Healthcare systems need to reorganize to provide high-quality care without increasing costs to an aging population with a high prevalence of chronic and long-term conditions. Several leading international health organizations, including the World Health Organization and the National Academy of Medicine, have emphasized the need to move toward increasingly person-centered healthcare systems. When healthcare is provided within the framework of Person-Centered Care (PCC), personal experiences, life stories, family, environment, and goals and desires are considered when planning health-related aspects. Each individual's subjectivity must be regarded as how they integrate into their environment and what their strengths and weaknesses, future plans, and rights are.

The SHARE study is expected to improve several key outcome indicators that enhance individuals' life experiences by combining current healthcare with the PCC approach. By reducing care demand, it will also contribute to the sustainability of the healthcare system.

Design This is an open-label, multicenter, randomized controlled clinical trial with parallel groups. It will be conducted as a superiority trial, where treatment comparisons will be made using "intention-to-treat" analysis. The study is based on the methodological framework of the Medical Research Council (MRC), which guides the development and evaluation of complex interventions. This research mainly focuses on studying effectiveness, i.e., to what extent the intervention achieves the intended outcomes in a real-world setting. The effect of a PCC intervention, in addition to the usual care received by individuals with CHF (intervention group), will be compared to usual care alone (control group).

Study setting / Context Outpatient Heart Failure Units at the OSI Donostialdea, the University Hospital of Navarra, and the University of Navarra Clinic in Pamplona.

Participants and recruitment procedure Participants will be recruited based on patient records from the CHF units at each hospital. The nursing professionals responsible for monitoring these patients, who will also be part of the research team, will review their weekly schedules and, using the described selection criteria, call potential participants a few days before their appointment to inform them about the possibility of participating in the study. On the day of the in-person consultation, the nurses will verbally explain the purpose of the study to the patients again and provide them with an information sheet for review. If they agree to participate, informed consent will be provided, and participants will be randomly assigned to the control or intervention group.

Study population The sample will consist of individuals with CHF who are being monitored for their condition at the hospitals mentioned above and meet the selection criteria.

Control group/Usual care These patients will not receive the intervention. Based on the European Society of Cardiology guidelines for managing these patients, they will receive the usual care for outpatient follow-up of their Chronic Heart Failure.

Intervention group In addition to standard care, patients in this group will receive the person-centered care intervention. They will have an initial in-person consultation (T0) with the nurse from the Heart Failure Unit. In this first session, the intervention will involve establishing a collaborative nurse-patient/family partnership, obtaining the patient's narrative, and designing and documenting a health plan. Through various communication skills, such as using open-ended questions, reflections, or summaries, the nurse will encourage the patient to share a narrative about their daily personal experiences and how CHF affects them, including the types of challenges they face and the resources available to them. During this dialogue, the nurse will take notes on the most relevant aspects of the narrative and identify the patient's health-related goals, capabilities, potential, personal/environmental resources, and needs. The patient (sometimes with their family) and the nurse will co-create a care plan collaboratively.

Additionally, the patient will be informed about scheduling a monthly phone appointment over the next three months with the same nurse to continue the plan and update the information related to the five elements recorded in the previous consultation, adapting them to new circumstances. The updated and agreed-upon plan will be sent to the patient's home by email or regular mail. Finally, the third-month consultation (T1) will serve to evaluate the last month's progress, plan longer-term goals with the patient, guide them in achieving these goals, and conclude the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals over 18 years old;
2. Functional class II-IV according to the NYHA;
3. Adequate cognitive status and health condition that allows participation;
4. Adequate spoken and written Spanish proficiency;
5. Active phone line; and
6. Voluntary signature of informed consent.

Exclusion Criteria:

1. Having a severe concurrent illness;
2. Life expectancy of less than 1 year;
3. Receiving palliative care;
4. Severe hearing impairment; and
5. Known alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of a PCC intervention on the ability to participate in social roles and activities in individuals with CHF. | Baseline, 3, 6 months.
  Neuro-QOL Item Bank v1.0 - Ability to Participate in Social Roles and Activities - Short Form A. (58). It consists of 7 items. Although originally designed for administration to individuals with chronic neurological conditions, this tool has been shown to be valid for use in other chronic conditions. It assesses the degree of participation in usual social roles, activities, and responsibilities, including work, family, friends, and leisure.
Evaluate the effect of a PCC intervention on perceived self-efficacy in individuals with CHF. | Baseline, 3, 6 months.
  General Self-Efficacy Scale (GSE) (60). This scale consists of 10 items and assesses the strength of an individual's belief in their own ability to respond to new or challenging situations and to overcome obstacles and setbacks.

SECONDARY OUTCOMES:
Evaluate the effect of a PCC intervention on the perceived level of social isolation in individuals with CHF. | Time Frame: Baseline, 3, 6 months.
  Revised UCLA Loneliness Scale (R-UCLA) (59). For this study, only the domain measuring social isolation, which contains 10 items, will be administered. This scale is designed to measure subjective feelings of loneliness as well as feelings of social isolation.
Evaluate the effect of a PCC intervention on the perceived social support in individuals with CHF. | Baseline, 3, 6 months.
  modified Medical Outcomes Study Social Support Survey (mMOS-SS) . This scale consist of items and is the abbreviated version of the MOS-SS scale designed to assess the perception of social support in people with chronic conditions. This version contains two subscales covering two domains, social/emotional and instrumental support.
Evaluate the effect of a PCC intervention on self-care behaviors in individuals with CHF. | Baseline, 3, 6 months.
  European Heart Failure Self-care Behaviour Scale (EHFScB-9) (63). This scale consists of 9 items and addresses aspects related to patient self-care behaviors, such as daily weight monitoring, fluid restriction, medication adherence, exercise, and contacting a healthcare professional.
Evaluate the effect of a PCC intervention on the experience of living with CHF. | Baseline, 3, 6 months.
  UNAV-Experience of Living with Chronic Heart Failure Scale (UNAV-CHF Experience Scale) (Olano-Lizarraga et al., in publication phase): This scale consists of 30 items and was designed to understand the experience of individuals living with CHF. It evaluates five dimensions: profound personal change, acceptance of the illness, perception of normality, hope, and perception of negatively impacting the family.
Evaluate the effect of a PCC intervention on the quality of life of individuals with CHF. | Baseline, 3, 6 months.
  Kansas City Cardiomyopathy Questionnaire (KCCQ): This scale consists of 23 items and assesses health-related quality of life in individuals with CHF. It evaluates seven domains: physical limitation; symptoms, considering changes over time, frequency, and severity; self-efficacy and knowledge; quality of life; and social interference.
Evaluate the effect of a PCC intervention on anxiety and depression levels in individuals with CHF. | Baseline, 3, 6 months.
  Hospital Anxiety and Depression Scale (HADS): This scale consists of 14 items, with 7 items in the anxiety subscale and 7 in the depression subscale. It was developed to indicate the possible presence of anxiety and depression in non-psychiatric outpatient patients.

OTHER OUTCOMES:
Evaluate the effect of a PCC intervention on hospitalization rates in individuals with CHF. | Baseline, 3, 6 months.
  Hospitalizations: The rate of unplanned hospitalizations related to CHF during the intervention and follow-up; data obtained from the medical record.
Evaluate the effect of a PCC intervention on decompensation rates in individuals with CHF. | Baseline, 3, 6 months.
  Decompensations: The rate of symptomatic CHF decompensations during the intervention and follow-up; data obtained from the medical record.
Evaluate the effect of a PCC intervention on the number of emergency department visits in individuals with CHF. | Baseline, 3, 6 months.
  Unscheduled visits: The number of unscheduled emergency department visits related to CHF; data obtained from the medical record.
Evaluate the effect of a PCC intervention on all-cause mortality in individuals with CHF. | Baseline, 3, 6 months.
  Death: Death from any cause; data obtained from the medical record.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Navarra, Facultad de Enfermería, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali L, Wallstrom S, Barenfeld E, Fors A, Fredholm E, Gyllensten H, Swedberg K, Ekman I. Person-centred care by a combined digital platform and structured telephone support for people with chronic obstructive pulmonary disease and/or chronic heart failure: study protocol for the PROTECT randomised controlled trial. BMJ Open. 2020 Jul 19;10(7):e036356. doi: 10.1136/bmjopen-2019-036356. PMID 32690519
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. Int J Nurs Stud. 2024 Jun;154:104705. doi: 10.1016/j.ijnurstu.2024.104705. Epub 2024 Feb 24. PMID 38564982
- [Background] Markgren R, Brannstrom M, Lundgren C, Boman K. Impacts of person-centred integrated chronic heart failure and palliative home care on pharmacological heart failure treatment: a substudy of a randomised trial. BMJ Support Palliat Care. 2019 Mar;9(1):e10. doi: 10.1136/bmjspcare-2015-000894. Epub 2016 Jan 20. PMID 26792391
- [Background] Brannstrom M, Boman K. Effects of person-centred and integrated chronic heart failure and palliative home care. PREFER: a randomized controlled study. Eur J Heart Fail. 2014 Oct;16(10):1142-51. doi: 10.1002/ejhf.151. Epub 2014 Aug 27. PMID 25159126
- [Background] Wallstrom S, Ali L, Ekman I, Swedberg K, Fors A. Effects of a person-centred telephone support on fatigue in people with chronic heart failure: Subgroup analysis of a randomised controlled trial. Eur J Cardiovasc Nurs. 2020 Jun;19(5):393-400. doi: 10.1177/1474515119891599. Epub 2019 Nov 29. PMID 31782661
- [Background] Fors A, Blanck E, Ali L, Ekberg-Jansson A, Fu M, Lindstrom Kjellberg I, Makitalo A, Swedberg K, Taft C, Ekman I. Effects of a person-centred telephone-support in patients with chronic obstructive pulmonary disease and/or chronic heart failure - A randomized controlled trial. PLoS One. 2018 Aug 31;13(8):e0203031. doi: 10.1371/journal.pone.0203031. eCollection 2018. PMID 30169539
- [Background] Ekman I, Wolf A, Olsson LE, Taft C, Dudas K, Schaufelberger M, Swedberg K. Effects of person-centred care in patients with chronic heart failure: the PCC-HF study. Eur Heart J. 2012 May;33(9):1112-9. doi: 10.1093/eurheartj/ehr306. Epub 2011 Sep 15. PMID 21926072
- [Background] Ekman I, Ebrahimi Z, Olaya Contreras P. Person-centred care: looking back, looking forward. Eur J Cardiovasc Nurs. 2021 Apr 13;20(2):93-95. doi: 10.1093/eurjcn/zvaa025. PMID 33693738
- [Background] Olano-Lizarraga M, Wallstrom S, Martin-Martin J, Wolf A. Interventions on the social dimension of people with chronic heart failure: a systematic review of randomized controlled trials. Eur J Cardiovasc Nurs. 2023 Mar 1;22(2):113-125. doi: 10.1093/eurjcn/zvac051. PMID 35737922
- [Background] Olano-Lizarraga M, Wallstrom S, Martin-Martin J, Wolf A. Causes, experiences and consequences of the impact of chronic heart failure on the person s social dimension: A scoping review. Health Soc Care Community. 2022 Jul;30(4):e842-e858. doi: 10.1111/hsc.13680. Epub 2021 Dec 16. PMID 34918403
- [Background] Olano-Lizarraga M, Martin-Martin J, Perez-Diez Del Corral M, Saracibar-Razquin M. Experiencing the possibility of near death on a daily basis: A phenomenological study of patients with chronic heart failure. Heart Lung. 2022 Jan-Feb;51:32-39. doi: 10.1016/j.hrtlng.2021.08.006. Epub 2021 Oct 29. PMID 34731695
- [Background] Olano-Lizarraga M, Zaragoza-Salcedo A, Martin-Martin J, Saracibar-Razquin M. Redefining a 'new normality': A hermeneutic phenomenological study of the experiences of patients with chronic heart failure. J Adv Nurs. 2020 Jan;76(1):275-286. doi: 10.1111/jan.14237. Epub 2019 Nov 4. PMID 31642086
- [Background] Olano-Lizarraga M, Oroviogoicoechea C, Errasti-Ibarrondo B, Saracibar-Razquin M. The personal experience of living with chronic heart failure: a qualitative meta-synthesis of the literature. J Clin Nurs. 2016 Sep;25(17-18):2413-29. doi: 10.1111/jocn.13285. Epub 2016 Jun 6. PMID 27273246
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Ekman I, Swedberg K, Taft C, Lindseth A, Norberg A, Brink E, Carlsson J, Dahlin-Ivanoff S, Johansson IL, Kjellgren K, Liden E, Ohlen J, Olsson LE, Rosen H, Rydmark M, Sunnerhagen KS. Person-centered care--ready for prime time. Eur J Cardiovasc Nurs. 2011 Dec;10(4):248-51. doi: 10.1016/j.ejcnurse.2011.06.008. Epub 2011 Jul 20. PMID 21764386